CLINICAL TRIAL: NCT03436849
Title: Phase 1 Study of ESN364 - Placebo-controlled, Single and Multiple Oral Dose Study in Healthy Japanese Male and Healthy Japanese Pre- and Postmenopausal Female Subjects -
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ESN364 in Healthy Japanese Male and Pre- and Post-menopausal Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2693-CL-0020
Record Dates: First submitted 2018-01-30; First posted 2018-02-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2019-04

CONDITIONS: Healthy Subjects
Keywords: ASP2693; Pharmacodynamics; Pharmacokinetics; ESN364; Safety
MeSH Terms: interventions — fezolinetant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- ESN364 dose-1 group in Part 1 (Experimental): Healthy male subjects will receive a single dose of ESN364.
  Interventions: Drug: ESN364
- ESN364 dose-2 group in Part 1 (Experimental): Healthy male subjects will receive a single dose of ESN364.
  Interventions: Drug: ESN364
- Placebo group in Part 1 (Placebo Comparator): Healthy male subjects will receive a single dose of Placebo.
  Interventions: Drug: Placebo
- Male ESN364 group in Part 2 (Experimental): Healthy male subjects will receive a single dose of ESN364 followed by washout period, then receive once daily dosing of ESN364 for 10 consecutive days at the same dose level.
  Interventions: Drug: ESN364
- Pre-menopausal female ESN364 group in Part 2 (Experimental): Healthy pre-menopausal female subjects will receive a single dose of ESN364 followed by washout period, then receive once daily dosing of ESN364 for 10 consecutive days at the same dose level.
  Interventions: Drug: ESN364
- Post-menopausal female ESN364 group in Part 2 (Experimental): Healthy post-menopausal female subjects will receive a single dose of ESN364 followed by washout period, then receive once daily dosing of ESN364 for 10 consecutive days at the same dose level.
  Interventions: Drug: ESN364
- Male placebo group in Part 2 (Placebo Comparator): Healthy male subjects will receive a single dose of Placebo followed by washout period, then receive once daily dosing of Placebo for 10 consecutive days.
  Interventions: Drug: Placebo
- Pre-menopausal female placebo group in Part 2 (Placebo Comparator): Healthy pre-menopausal female subjects will receive a single dose of Placebo followed by washout period, then receive once daily dosing of Placebo for 10 consecutive days.
  Interventions: Drug: Placebo
- Post-menopausal female placebo group in Part 2 (Placebo Comparator): Healthy post-menopausal female subjects will receive a single dose of Placebo followed by washout period, then receive once daily dosing of Placebo for 10 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ESN364 — ESN364 will be administered orally.
  Arms: ESN364 dose-1 group in Part 1; ESN364 dose-2 group in Part 1; Male ESN364 group in Part 2; Post-menopausal female ESN364 group in Part 2; Pre-menopausal female ESN364 group in Part 2
Drug: Placebo — Placebo will be administered orally.
  Arms: Male placebo group in Part 2; Placebo group in Part 1; Post-menopausal female placebo group in Part 2; Pre-menopausal female placebo group in Part 2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple oral doses of ESN364 in healthy Japanese male and pre- and post-menopausal female subjects. This study will also evaluate the pharmacokinetics (PK) of ESN364 and its metabolite, and the pharmacodynamics (PD) of ESN364 after single and multiple oral doses administration in healthy Japanese male and pre- and post-menopausal female subjects.

DETAILED DESCRIPTION:
This study consists of two parts. Part 1; Single Dose (SD) and Part 2; Single and Multiple Dose (SD and MD).

ELIGIBILITY:
Inclusion Criteria:

* Male subject between 20 to < 45 years of age, or female subject between 20 to < 65 years of age.
* Body weight at screening: ≥ 50.0 kg and < 80.0 kg for male, ≥ 40.0 kg and < 70.0 kg for female.
* Body mass index (BMI) at screening: range of ≥ 17.6 kg/m2 and < 26.4 kg/m2 [BMI = Body weight (kg) ÷ {Body height (m)2}].

Exclusion Criteria:

* Subjects who participated or are scheduled to participate in any clinical trials or post-marketing studies within 84 days prior to screening.
* Subject has had previous exposure with ESN364.
* Subject has any clinically significant history of allergic conditions prior to study drug administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy.
* Subject has contracted pyretic or symptomatic viral, bacterial, or fungal infection within 7 days prior to hospital admission.
* Any deviation from the normal range of blood pressure, pulse, body temperature, or routine 12-lead ECG at screening or on the day of hospital admission.
* Subjects who has any significantly abnormal results of laboratory tests at screening or on the day of hospital admission.
* Subjects who are positive for any of urinary drug abuse test or serology test at screening.
* Subject took a drug or underwent therapy within 2 weeks prior to hospital admission.
* Subjects used a drug or underwent therapy that affects sex hormones within 3 months prior to hospital admission.
* Subjects who had bilateral orchiectomy.
* Subject has used any inducer of metabolism in the 3 months prior to hospital admission.
* Subject has a history of smoking more than 10 cigarettes per day within 3 months prior to screening test.
* Subject consumes, on average, more than approximately 500 mg/day of caffeine
* Subject has a history of consuming more than 30 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/ substance abuse within past 2 years prior to screening.
* Subjects who conducted or is scheduled to conduct any blood donation or blood drawing.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of adverse events (AEs) in Part 1 | Up to Day 12 in Part 1
  AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA).
Safety assessed by incidence of AEs in Part 2 | Up to Day 24 in Part 2
  AEs will be coded using MedDRA.
Safety assessed by vital signs: Body temperature in Part 1 | Up to day 12 in Part 1
  To assess vital signs as a criterion of safety variables.
Safety assessed by vital signs: Body temperature in Part 2 | Up to Day 24 in Part 2
  To assess vital signs as a criterion of safety variables.
Safety assessed by vital signs: Blood pressure in Part 1 | Up to Day 12 in Part 1
  To assess vital signs as a criterion of safety variables.
Safety assessed by vital signs: Blood pressure in Part 2 | Up to Day 24 in Part 2
  To assess vital signs as a criterion of safety variables.
Safety assessed by vital signs: Pulse rate in Part 1 | Up to Day 12 in Part 1
  To assess vital signs as a criterion of safety variables.
Safety assessed by vital signs: Pulse rate in Part 2 | Up to Day 24 in Part 2
  To assess vital signs as a criterion of safety variables.
Safety assessed by laboratory test: Hematology in Part 1 | Up to Day 12 in Part 1
  To assess laboratory values as a criterion of safety variables. Potentially clinically significant laboratory values will be reported as AEs.
Safety assessed by laboratory test: Hematology in Part 2 | Up to Day 24 in Part 2
  To assess laboratory values as a criterion of safety variables. Potentially clinically significant laboratory values will be reported as AEs.
Safety assessed by laboratory test: Biochemistry in Part 1 | Up to Day 12 in Part 1
  To assess laboratory values as a criterion of safety variables. Potentially clinically significant laboratory values will be reported as AEs.
Safety assessed by laboratory test: Biochemistry in Part 2 | Up to Day 24 in Part 2
  To assess laboratory values as a criterion of safety variables. Potentially clinically significant laboratory values will be reported as AEs.
Safety assessed by laboratory test: Urinalysis in Part 1 | Up to Day 12 in Part 1
  To assess laboratory values as a criterion of safety variables. Potentially clinically significant laboratory values will be reported as AEs.
Safety assessed by laboratory test: Urinalysis in Part 2 | Up to Day 24 in Part 2
  To assess laboratory values as a criterion of safety variables. Potentially clinically significant laboratory values will be reported as AEs.
Safety assessed by standard 12-lead electrocardiogram (ECG) in Part 1 | Up to Day 12 in Part 1
  Subjects should keep rest for 5 minutes before evaluation. Any clinically significant adverse changes on the ECG will be reported as AEs.
Safety assessed by standard ECG in Part 2 | Up to Day 24 in Part 2
  Subjects should keep rest for 5 minutes before evaluation. Any clinically significant adverse changes on the ECG will be reported as AEs.
Safety assessed by ECG parameters: Heart rate in Part 1 | Up to 24 hr after dosing in Part 1
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: Heart rate in Part 2 | Up to 24 hr after dosing on Day 10 in multiple dose (MD) of Part 2
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: QT interval in Part 1 | Up to 24 hr after dosing in Part 1
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: QT interval in Part 2 | Up to 24 hr after dosing on Day 10 in MD of Part 2
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: RR interval in Part 1 | Up to 24 hr after dosing in Part 1
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: RR interval in Part 2 | Up to 24 hr after dosing on Day 10 in MD of Part 2
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: PR interval in Part 1 | Up to 24 hr after dosing in Part 1
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: PR interval in Part 2 | Up to 24 hr after dosing on Day 10 in MD of Part 2
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: QRS interval in Part 1 | Up to 24 hr after dosing in Part 1
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: QRS interval in Part 2 | Up to 24 hr after dosing on Day 10 in MD of Part 2
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: QTc interval corrected by Fridericia method (QTcF) in Part 1 | Up to 24 hr after dosing in Part 1
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by ECG parameters: QTcF in Part 2 | Up to 24 hr after dosing on Day 10 in MD of Part 2
  To assess ECG parameters as a criterion of safety variables.
Safety assessed by body weight in Part 1 | Up to Day 3 in Part 1
  To assess body weight as a criterion of safety variables
Safety assessed by body weight in Part 2 | Up to Day 15 in Part 2
  To assess body weight as a criterion of safety variables
Safety assessed by menstrual cycle in pre-menopausal females | Up to an average of two weeks after last dosing
  To assess menstrual cycle as a criterion of safety variables

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter for ESN364 and its metabolite: Area under the concentration-time curve (AUC) from the time of dosing to time 24 h (AUC24) in plasma | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2
  To assess the PK of ESN364 and its metabolite in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: AUC from the time of dosing extrapolated to time infinity (AUCinf) in plasma | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2
  To assess the PK of ESN364 and its metabolite4 in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: Percentage of AUCinf (AUCinf(%extrap)) in plasma | Up to 48 hr after dosing in Part 1
  To assess the PK of ESN364 and its metabolite in Part 1.
PK parameter for ESN364 and its metabolite: AUC from the time of dosing to the last measurable concentration (AUClast) in plasma | Up to 48 hr after dosing in Part 1
  To assess the PK of ESN364 and its metabolite in Part 1.
PK parameter for ESN364 and its metabolite: Maximum concentration (Cmax) in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: Apparent total clearance after extra-vascular dosing (CL/F) in plasma | Up to 48 hr after dosing in Part 1 and after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: Time point prior to the time point corresponding to the first measurable (non-zero) concentration (tlag) in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: Time of the maximum concentration： (tmax) in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: Terminal elimination half-life (t1/2) in plasma | Up to 48 hr after dosing in Part 1 and after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: volume of distribution during the terminal elimination phase after extra-vascular dosing (Vz/F) in plasma | Up to 48 hr after dosing in Part 1 and after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 1 and Part 2.
PK parameter for ESN364 metabolite: Metabolite to parent ratio (MPR) in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 metabolite in Part 1 and Part 2.
PK parameter for ESN364 and its metabolite: AUC from the time of dosing to the start of the next dosing interval (AUCtau) in plasma | Up to 48 hr after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 2.
PK parameter for ESN364 and its metabolite: Peak-trough ratio (PTR) in plasma | Up to 48 hr after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 2.
PK parameter for ESN364 and its metabolite: Accumulation ratio calculated using AUC (Rac(AUC)) in plasma | Up to 48 hr after dosing on Day 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 2.
PK parameter for ESN364 and its metabolite: Concentration immediately prior to dosing at multiple dosing (Ctrough) in plasma | Before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PK of ESN364 and its metabolite in Part 2.
Pharmacodynamic (PD) endpoint for ESN364: Luteinizing hormone (LH) level in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC12 for LH level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC24 for LH level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC48 for LH level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Cmin for LH level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: tmin for LH level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC from the Time of Dosing to the Start of the Next Dosing Interval (AUCtau) for LH level | Before dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 2.
PD endpoint for ESN364: Cpredose for LH level | Before dosing in Part 1 and before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Follicle stimulating hormone (FSH) level in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC12 for FSH level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC24 for FSH level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC48 for FSH level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Cmin for FSH level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: tmin for FSH level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUCtau for FSH level | Before dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 2.
PD endpoint for ESN364: Cpredose for FSH level | Before dosing in Part 1 and before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Sex hormone binding globulin (SHBG) level in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC12 for SHBG level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC24 for SHBG level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC48 for SHBG level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Cmin for SHBG level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: tmin for SHBG level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUCtau for SHBG level | Before dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 2.
PD endpoint for ESN364: Cpredose for SHBG level | Before dosing in Part 1 and before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Total testosterone (TT) level in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC24 for TT level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC12 for TT level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC48 for TT level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Cmin for TT level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: tmin for TT level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUCtau for TT level | Before dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 2.
PD endpoint for ESN364: Cpredose for TT level | Before dosing in Part 1 and before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Free testosterone (FT) level in plasma | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC12 for FT level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC24 for FT level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUC48 for FT level | Up to 48 hr after dosing in Part 1 and after first dosing in Part 2.
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Cmin for FT level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: tmin for FT level | Up to 48 hr after dosing in Part 1, after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: AUCtau for FT level | Before dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 2.
PD endpoint for ESN364: Cpredose for FT level | Before dosing in Part 1 and before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PD of ESN364 in Part 1 and Part 2.
PD endpoint for ESN364: Estradiol (E) level in plasma | Up to 48 hr after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUC12 for E level | Up to 48 hr after first dosing in Part 2.
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUC24 for E level | Up to 48 hr after first dosing in Part 2.
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUC48 for E level | Up to 48 hr after first dosing in Part 2.
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: Cmin for E level | Up to 48 hr after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: tmin for E level | Up to 48 hr after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUCtau for E level | Before dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: Cpredose for E level | Before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: Progesterone (P) level in plasma | Up to 48 hr after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUC12 for P level | Up to 48 hr after first dosing in Part 2.
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUC24 for P level | Up to 48 hr after first dosing in Part 2.
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUC48 for P level | Up to 48 hr after first dosing in Part 2.
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: Cmin for P level | Up to 48 hr after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: tmin for P level | Up to 48 hr after first dosing in Part 2 and after dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: AUCtau for P level | Before dosing on Day 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.
PD endpoint for ESN364: Cpredose for P level | Before dosing on Day 2, 3, 5, 7 and 10 in MD part of Part 2
  To assess the PD of ESN364 in female subjects in Part 2.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.